CLINICAL TRIAL: NCT00708981
Title: Combined Diabetes-Renal Multifactorial Intervention In Patients With Advanced Diabetic Nephropathy (ADN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook County Health (Other Government)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Leon Fogelfeld MD, M.D., Cook County Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-177 Metabolism IST; IRB 06-177 (Other: John H Stroger Hospital IRB)
Record Dates: First submitted 2008-06-26; First posted 2008-07-03 (Estimated); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Active Comparator): Study group will receive multifactorial intervention for advanced diabetic nephropathy:
  Elements of multifactorial intervention:
  1. BP control of <130/80mmHg and renal protection with reduction of proteinuria to <0.5g/day using therapy with ACE inhibitors and/or ARBs.
  2. Tight glucose control with target of HbA1C of 7% and below using SMBG and Lantus/Apidra regimen.
  3. Use of hypolipidemic therapy to achieve targets of LDL < 70 mg/dl, HDL > 40/50 mg/dl (M/F)and TG < 200 mg/dl.
  4. Patient enhanced self-management provided by combined diabetes-renal education curriculum.
  5. Behavior and social intervention
  6. Intense case management that includes close follow-up of visits, laboratory monitoring and other self-adherence behaviors carried out by clinical research coordinators.
  Interventions: Other: Multifactorial Intervention
- Control Group (No Intervention): Control Group will keep on receiving the usual treatment that they used to receive from their respective clinics and the Diabetes-Renal team would not alter their therapy or interfere in their management.

INTERVENTIONS:
Other: Multifactorial Intervention — Study group will receive multifactorial intervention for advanced diabetic nephropathy:
  Elements of multifactorial intervention:
  1. BP control of <130/80mmHg and renal protection with reduction of proteinuria to <0.5g/day using therapy with ACE inhibitors and/or ARBs.
  2. Tight glucose control with target of HbA1C of 7% and below using SMBG and Lantus/Apidra regimen.
  3. Use of hypolipidemic therapy to achieve targets of LDL < 70 mg/dl, HDL > 40/50 mg/dl (M/F)and TG < 200 mg/dl.
  4. Patient enhanced self-management provided by combined diabetes-renal education curriculum.
  5. Behavior and social intervention
  6. Intense case management that includes close follow-up of visits, laboratory monitoring and other self-adherence behaviors carried out by clinical research coordinators.
  Arms: Study Group

SUMMARY:
The purpose of this study is to compare the progression of kidney disease in subjects with Diabetes mellitus type 2 and Advanced Diabetic Nephropathy treated by routine follow-up as a general care and in subjects treated by multi-factorial intervention in the Diabetes-Renal Clinic.

DETAILED DESCRIPTION:
In this study, the overall objective is comparison of progression of renal insufficiency in subjects with Advanced Diabetic Nephropathy (CKD stages 3 and 4) randomized into multifactorial intervention in the Diabetes-Renal Clinic (study group) and into usual care (control group). The multifactorial intervention includes the following: 1. Blood pressure control to the goal of <130/80mmHg and renal protection with reduction of proteinuria to <0.5g/day using a protocol that includes therapy with ACE inhibitors, ARBs or their combination. 2. Tight glucose control using SMBG and Lantus/Apidra self-escalation regimen. 3. Use of hypolipidemic therapy to achieve targets of LDL of < 70 mg/dl, HDL > 40/50 mg/dl (males/females) [since you said that HDL is not a target because there are no meds for it I deleted HDL;] and triglycerides of less than 200 mg/dl. 4. Patient enhanced self-management provided by combined diabetes-renal education curriculum (taught by certified diabetes and renal educators). 5. Behavior and social intervention (motivational interviews and social assessment) provided as needed by social workers. 6. Intense case management that includes close follow-up of visits, laboratory monitoring and other self-adherence behaviors. 7. Weight loss with lifestyle and diet modification.

Control Group will keep on receiving the usual treatment that they used to receive from their respective clinics and the Diabetes-Renal team would not alter their therapy or interfere in their management.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is male or female diagnosed with Type 2 Diabetes mellitus defined by the American Diabetes Association criteria and must be aged 18 to 70 years.
2. The participant must have documented Advanced Diabetic Nephropathy (ADN) defined as presence of proteinuria or micro/macro-albuminuria and impaired GFR (by MDRD equation) corresponding to Chronic Kidney Disease (CKD) stages 3-4 (moderate-severe i.e. estimated GFR >15ml/min and <60ml/min).

   A. Presence of macroalbuminuria B. Presence of microalbuminuria if no therapy with ACE inhibitors or ARBs C. Presence of current microalbuminuria and previous documentation of macroalbuminuria D. Presence of current microalbuminuria and previous documentation of Diabetic Retinopathy or laser therapy E. If only microalbuminuria and no A, B, C or D US of kidney shows NL size.
3. Minimal cognitive function for a diabetes self management
4. Fasting or random Blood glucose <400mg/DL

Exclusion Criteria:

1. Patients with Type 1 Diabetes Mellitus.
2. Serum Creatinine > 4.0 mg/dl and/or an estimated GFR of < 15 ml/min.
3. Patients on renal replacement therapy.
4. Patients with Hyperkalemia (K>5.0 meq/L).
5. Patients with known Renal Artery stenosis.
6. Patients with known cancer, hepatic impairment, dementia or other chronic medical diseases.
7. Patients with severe heart failure (NYHA Class III or IV symptoms and/or LVEF <25%).
8. Patients with valvular or outflow tract obstruction.
9. Patients with significant disability that precludes regular attendance at clinics for follow-up.
10. Patients unwilling or unable to provide informed consent.
11. Pregnant or lactating women.
12. Current addiction to substance or alcohol abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-05; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Delay in development in end-stage renal failure in subjects with Advanced Diabetic Nephropathy (CKD stages 3 and 4) | 2 years
  Time to reaching End Stage Renal Disease (ESRD)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Fogelfeld, MD, Principal Investigator — John H. Stroger, Jr. Hospital of Cook County, Endocrinology
Locations (1):
- John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois, United States

REFERENCES:
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639